CLINICAL TRIAL: NCT03088462
Title: LiveWell: A Mobile Intervention for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Evan Goulding, Assistant Professor, Department of Psychiatry and Behavioral Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH110626 (NIH); 1R01MH110626 (NIH)
Record Dates: First submitted 2017-03-08; First posted 2017-03-23 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder; Bipolar I Disorder
Keywords: Bipolar Disorder; Smartphone; Behavior Therapy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Active Comparator): Any treatment for bipolar disorder participant is involved in.
  Interventions: Other: Psychiatric management; Behavioral: Psychosocial treatment
- Treatment As Usual + LiveWell Program (Experimental): Treatment as usual combined with the LiveWell program.
  Interventions: Other: Psychiatric management; Behavioral: Psychosocial treatment; Behavioral: LiveWell Program

INTERVENTIONS:
Other: Psychiatric management — Routine treatment for bipolar disorder with a psychiatrist including prescription of medications and potentially other treatments such as individual, group or light therapy.
Behavioral: Psychosocial treatment — Any psychosocial treatment participant is involved in such as individual therapy, group therapy, or support groups.
Behavioral: LiveWell Program — Participants work with a health coach to facilitate use of a smartphone application designed for people with bipolar disorder.
  Arms: Treatment As Usual + LiveWell Program

SUMMARY:
LiveWell is a study evaluating the use of smartphones to better understand and improve the treatment of bipolar disorder. Our goal is to increase access to psychosocial interventions and improve their effectiveness in reducing symptoms and preventing mood episodes.

DETAILED DESCRIPTION:
A single blind, randomized controlled trial (N = 200, 2:3 ratio of usual care vs usual care and intervention) will be conducted in clinical practices around Chicago and Minneapolis. Eligible participants are adult bipolar 1 disorder patients not experiencing a current mood episode with a history of at least one acute episode in the last two years who are in treatment with a psychiatrist.

The primary clinical outcome will be time to relapse, and the secondary outcomes will be percent time symptomatic, symptom severity, and quality of life.

Participation in the study lasts for 12 months. Participants are asked to carry a smartphone with them whenever they leave home and wear a wristwatch for measuring activity all day every day. Participants are also asked to complete a series of telephone assessments and may be asked to complete daily check-ins on a smartphone and work with a health coach.

Participants will need to attend two in-person clinic visits at 680 N Lake Shore Drive, Chicago IL 60611 Suite 1520 or at 3311 E Old Shakopee Rd, Bloomington, MN 55425.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years
* Bipolar Disorder Type I
* Minimum of 1 acute episode in the last 2 years

Exclusion Criteria:

* Not receiving psychiatric care
* Current mood episode
* Current substance use disorder (within the last 3 months)
* Current severe suicidal ideation or a recent serious suicide attempt (within the last 3 months)
* Inability to speak and read English
* Visual, hearing, voice, cognitive or motor impairment that would prevent completion of study and treatment procedures

Participants will need to attend two in-person clinic visits at 680 N Lake Shore Drive, Chicago IL 60611 Suite 1520 or at 3311 E Old Shakopee Rd, Bloomington, MN 55425.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Longitudinal Interval Follow-up Evaluation-Clinical Monitoring Form: Clinical Status | Up to 48 weeks
  Semi-structured interview designed to assess clinical status allowing determination of time to relapse (onset of a mood episode).
  Clinical Status: episode = depression, mania, hypomania, mixed; continued symptomatic (≥ 3 moderate symptoms without recovery), recovering (≤ 2 moderate symptoms, ≤ 8 weeks), prodromal (≥ 3 moderate symptoms after recovery); recovered (≤ 2 moderate symptoms, ≥ 8 weeks).

SECONDARY OUTCOMES:
Longitudinal Interval Follow-up Evaluation-Clinical Monitoring Form: Symptom Severity | 48 weeks
  Semi-structured interview designed to assess symptom severity allowing determination of percent time symptomatic (time with psychiatric status rating > 1.5).
  Psychiatric Status Rating: Syndromal Symptoms - 6 = definite criteria with psychotic symptoms or extreme impairment, 5 = definite criteria without psychotic symptoms or extreme impairment; Subsyndromal Symptoms - 4 = not definite criteria but major symptoms or major impairment, 3 = ≥ 3 moderate symptoms, moderate impairment, 2 = ≤ 2 moderate criteria symptoms, minimal impairment; Asymptomatic:1.5 = ≥ 1 mild but no moderate criteria symptoms; 1 = no mild or moderate criteria symptoms.
Change in Quick Inventory of Depressive Symptomatology-Clinician Rating | At 0, 8, 16, 24, 32, 40 and 48 weeks
  Structured interview designed to assess severity of depression. Scale range is from 0-27.
Change in Young Mania Rating Scale | At 0, 8, 16, 24, 32, 40 and 48 weeks
  Structured interview designed to assess severity of mania. Scale range is from 0-60.
Change in World Health Organization Quality of Life Scale (BREF) | At 0, 24 and 48 weeks
  Structured interview designed to assess physical health, psychological health, social relationships, and environment. Each domain is scored individually with transformed scores of 4-20.

CONTACTS AND LOCATIONS:
Overall Officials: Evan H Goulding, MD/PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - HealthPartners Institute, Bloomington, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jonathan GK, Abitante G, McBride A, Bernstein-Sandler M, Babington P, Dopke CA, Rossom RC, Mohr DC, Goulding EH. LiveWell, a smartphone-based self-management intervention for bipolar disorder: Intervention participation and usability analysis. J Affect Disord. 2024 Apr 1;350:926-936. doi: 10.1016/j.jad.2024.01.099. Epub 2024 Jan 19. PMID 38246280
- [Derived] Goulding EH, Dopke CA, Rossom R, Jonathan G, Mohr D, Kwasny MJ. Effects of a Smartphone-Based Self-management Intervention for Individuals With Bipolar Disorder on Relapse, Symptom Burden, and Quality of Life: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Feb 1;80(2):109-118. doi: 10.1001/jamapsychiatry.2022.4304. PMID 36542401
- [Derived] Goulding EH, Dopke CA, Rossom RC, Michaels T, Martin CR, Ryan C, Jonathan G, McBride A, Babington P, Bernstein M, Bank A, Garborg CS, Dinh JM, Begale M, Kwasny MJ, Mohr DC. A Smartphone-Based Self-management Intervention for Individuals With Bipolar Disorder (LiveWell): Empirical and Theoretical Framework, Intervention Design, and Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Feb 21;11(2):e30710. doi: 10.2196/30710. PMID 35188473